CLINICAL TRIAL: NCT04134052
Title: Effect of Regional Anesthesia and Sedation With Ketamine Versus Regional Anesthesia and Sedation With Midazolam in Cognitive Function in Patients Over 60 Years of Age in Elective Surgery at 3 Months of Postoperative Follow-up
Brief Title: Ketamine vs Midazolam on Cognitive Function in Elderly in Elective Surgery Three-Months Postoperatively (ketaminvsMDZ)
Acronym: ketaminvsMDZ
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Colima (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Pedro Julian Flores Moreno, Principal investigator, master of medical sciences, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 090129
Record Dates: First submitted 2019-10-05; First posted 2019-10-21 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Cognitive Dysfunction
Keywords: ketamine; midazolam; cognitive dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Simple finite randomization will be performed. The anesthesiologist will choose an envelope with an assigned folio divided into two groups 1) intravenous infusion midazolam and 2) intravenous infusion ketamine, For sedation, regional anesthesia will be applied and hemodynamic variables, administered drugs, type of surgery, surgery time and transoperative bleeding will be recorded, after that, the cognitive evolution will be evaluated with the minimental examination at 3 months postoperatively
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the participant, the researcher and the outcomes assesor don't know the drug used for sedation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ketamine sedation (Experimental): Sedation will be performed with ketamine dose 5-20mcg / kg / min in infusion with 100 ml Na Cl solution 0.9% during surgery
  Interventions: Drug: ketamine sedation versus midazolam sedation
- midazolam sedation (Active Comparator): Sedation will be performed with midazolam dose 5 - 35mcg / kg / hr in infusion with 100 ml Na Cl solution 0.9% during surgery
  Interventions: Drug: ketamine sedation versus midazolam sedation

INTERVENTIONS:
Drug: ketamine sedation versus midazolam sedation — Sedation with ketamine 5-20 mcg / kg / hr in infusion in 100ml Na Cl solution 0.9% during surgery and the second midazolam group 5 mcg- 35 mcg / kg / hr in infusion in 100ml Na Cl solution 0.9% will be administered during surgery
  Other Names: ketamine sedation

SUMMARY:
Deterioration of posoperative cognitive function (DCPO) is an intermediate state between normal cognitive aging and dementia, defined as a cognitive alteration greater than expected for the patient's age and educational level, but which doesn't interfere with the activities of daily life, in its evolution it can lead to dementia or it can present reversal of the deterioration with return to a normal cognitive state, or a stabilization with permanence in a state of moderate alteration. In general, higher cognitive function can be affected by organic or functional problems, anesthetic-surgical, diseases associated with the elderly and / or chronic-degenerative comorbidities. Older patients who undergo regional anesthesia have special interest, the adverse cardiovascular effects, or prolonged sedation due to a pharmacokinetics that is altered by age, call special attention to reduce complications in the postoperative period. In 2010 at the Siglo XXI Hospital in Mexico City, the 68-year-old population attended was 30% of those with postoperative cognitive dysfunction 26% a week, and 10% persistence at 3 months. The DSM V recommends a neuropsychiatric, psychological and cognitive evaluation of the patient in the postoperative period, through tests such as the Mini Mental State Examination. sub-anesthetic doses of ketamine have been recently proposed to reduce the postoperative markers of inflammation, pain and opioids, in addition to having an antidepressant effect. There is a pharmacological rationale for using ketamine as a preventative measure against postoperative delirium based on its N-methyl-D-aspartate (NMDA) antagonism, It has the potential to protect against such neurological injury.

DETAILED DESCRIPTION:
Randomized double blind clinical trial. Male and female patients 60-90 years of age scheduled in elective surgery under regional anesthesia and sedation.

The researchers will be double blind and the data analyzer will ignore the drug used ( it it should be midazolam or ketamine in an intravenous infusion). The principal investigator will limit himself to collecting the questionnaires and following up to 3 months. Simple finite randomization in two groups, will be done through envelopes.

The pre-surgical, post-surgical Mini Mental questionnaire will be applied on the first day, 1 month and 3 months. During the trans-anesthetic, hemodynamic variables and anesthetic depth index measurements will be taken, surgical time, estimated bleeding, use of other adjuvant medications, type of surgery and comorbidities will be taken as intervening variables.

ELIGIBILITY:
Inclusion Criteria:

* age 60-90 years,
* complete primary,
* ASA I-II,
* scheduled for non-urgent surgery,
* to whom regional anesthesia and sedation are applied
* sign the informed consent
* Able to answer the brief examination of the mental state (MMSE ) preliminary with more than 24 points

Exclusion Criteria:

* not able to respond to MMSE, deaf-mute, blindness,
* history of surgery the last 6 months,
* use of pacemakers,
* allergy to anesthetics,
* use of psychiatric medication, or drugs,
* diagnosed neurological disease (cerebrovascular disease, dementia, seizures) ,
* surgery scheduled for prostate resection, or reduction of hip fractures

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-01-24 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
cognitive function at baseline | It takes 30 minutes before the preparation of the surgery
  the mini mental examination test will be done at baseline for the diagnostic
Change the cognitive function #1 | It Will be done at the hospital after one day of recovery
  The minimental examination test Will be done after one day of the anesthesic procedure.
Change the cognitive function #2 | It Will be done at the patient home
  The minimental examination test Will be done after one month of the anesthesic procedure.
Change the cognitive function#3 | It Will be done at the patient home three months after the surgery
  The minimental examination test Will be done after three months of the anesthesic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar-Alberto Newton-Sanchez, Phd, Study Director — Universidad de Colima; Fabian Rojas-Larios, Phd, Principal Investigator — Universidad de Colima
Locations (1):
- Mexican Social Security Institute. General Hospital of Zone 1 Villa de Alvarez, Colima, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hogue CW, Grafman J. Aligning nomenclature for cognitive changes associated with anaesthesia and surgery with broader diagnostic classifications of non-surgical populations: a needed first step. Br J Anaesth. 2018 Nov;121(5):991-993. doi: 10.1016/j.bja.2017.12.029. Epub 2018 Jan 17. No abstract available. PMID 30336869
- [Result] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844
- [Result] Shoair OA, Grasso Ii MP, Lahaye LA, Daniel R, Biddle CJ, Slattum PW. Incidence and risk factors for postoperative cognitive dysfunction in older adults undergoing major noncardiac surgery: A prospective study. J Anaesthesiol Clin Pharmacol. 2015 Jan-Mar;31(1):30-6. doi: 10.4103/0970-9185.150530. PMID 25788770
- [Result] Li L, Vlisides PE. Ketamine: 50 Years of Modulating the Mind. Front Hum Neurosci. 2016 Nov 29;10:612. doi: 10.3389/fnhum.2016.00612. eCollection 2016. PMID 27965560
- [Result] Paredes S, Cortinez L, Contreras V, Silbert B. Post-operative cognitive dysfunction at 3 months in adults after non-cardiac surgery: a qualitative systematic review. Acta Anaesthesiol Scand. 2016 Sep;60(8):1043-58. doi: 10.1111/aas.12724. Epub 2016 Mar 29. PMID 27027720